CLINICAL TRIAL: NCT05930652
Title: Impact of Cumulative Stress on Mental Health in Young Adults
Brief Title: Cumulative Stress and Mental Health in Young Adults
Status: Completed | Type: Observational
Sponsor: Bernadetta Izydorczyk (Other)
Collaborators: Jagiellonian University (Other)
Responsible Party: Sponsor-Investigator, Bernadetta Izydorczyk, Professor, Jagiellonian University
Organization: Jagiellonian University (Other)
Other Study IDs: 221.0042.26_2023
Record Dates: First submitted 2023-06-26; First posted 2023-07-05 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-06

CONDITIONS: Stress, Psychological; Stress-related Problem; Cumulative Trauma; Mental Health Issue; Mental Stress; Psychological Well-Being
Keywords: cumulative stress; mental health; young adults; stress syndrome; risk factors; protective factors
MeSH Terms: conditions — Stress, Psychological; Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Young adults: The population of Polish Students, who graduated from high schools/ passed leaving exams, started university studies between 2020 and 2023, and were living in Poland during this period (2020-2023: COVID-19, lockdown, economic crisis, political changes, climate changes, and the war in Ukraine).
  Interventions: Diagnostic Test: Psychological tests and psychosocial questionnaires

INTERVENTIONS:
Diagnostic Test: Psychological tests and psychosocial questionnaires — Assessment of psychological functioning (including well-being, mental health conditions, coping skills), and socio-demographics, academic performance, home, relationships, general health, habits, and attitudes.

SUMMARY:
The goal of this observational study is to learn about the needs of young adults - "policrisis generation", exposed to cumulative stress during 2020-2023, in terms of quality of mental health, the psychosocial resources, protective factors for cumulative stress effect, and the standards for effective prevention. The main questions to be answered are:

* How does cumulative stress affect young adults?
* Is there a specific cumulative stress syndrome that can be described?
* What are the risk and the protective factors for cumulative stress?
* How does the "policrisis generation" deal with the cumulative stress they have been exposed to? Participants will complete psychological questionnaires

DETAILED DESCRIPTION:
Background: Epidemiological data are not sufficient to determine the mental health outcomes of exposure to cumulative stress of 2020-2023. Holistic knowledge of risk and protective factors, pathways leading to symptoms (not yet observed), and stress management strategies for the generation living under cumulative stress conditions (pandemic, war, refugee migration, economic crisis) is needed.

Participants: 400 young adults, recruited among university students.

Research methodology: Analysis of data collected by screening questionnaires, psychological scales, and questionnaires, related to mental health conditions.

ELIGIBILITY:
Inclusion Criteria:

* Age between 19 and 25 years
* Standard educational opportunities
* Attending the university course cycle

Exclusion Criteria:

* Age below 19
* Intellectual disability
* Inability to self-complete the research questionnaires

Ages: 19 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: University students participating in active learning.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2023-04-12 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
General Well-being | April 12, 2023 until June 15, 2023
  Global Flourishing Study Questionnaire Development Report (GFS). The GFS includes 12 questions that gauge respondents' level of "flourishing" across six domains: (1) happiness and life satisfaction, (2) mental and physical health, (3) meaning and purpose, (4) character and virtue, (5) close social relationships and (6) financial and material stability.
Personality Traits | April 12, 2023 until June 15, 2023
  Personality Inventory for ICD-11 (PiCD). The four-factor structure of the Polish version of PiCD consists of three unipolar factors as Negative Affectivity, Detachment, and Dissociality factors, and one bipolar Anankastia vs. Disinhibition factor.
Emotion Regulation | April 12, 2023 until June 15, 2023
  The Difficulties in Emotion Regulation Scale (DERS). It comprises the following dimensions: (1) lack of acceptance of emotional responses, (2) difficulties in realizing goal-directed behaviors, (3) difficulties in controlling impulses, (4) lack of emotional awareness, (5) limited access to emotion regulation strategies, (6) lack of emotional clarity
Meaning in Life | April 12, 2023 until June 15, 2023
  Meaning in Life Questionnaire (MLQ). A 10-item questionnaire designed to measure two dimensions of meaning in life: (1) Presence of Meaning (how much respondents feel their lives have meaning), and (2) Search for Meaning (how much respondents strive to find meaning and understanding in their lives).

SECONDARY OUTCOMES:
Authors survey | April 12, 2023 until June 15, 2023
  Survey of socio-demographic data (gender, age, sexual orientation, marital status, family, relationships, socio-economic status, place of residence, educational level, habits, attitudes, others)

CONTACTS AND LOCATIONS:
Overall Officials: Bernadetta Izydorczyk, Prof, Principal Investigator — Institute of Psychology, Jagiellonian University in Krakow, 30-060 Krakow, Poland
Locations (1):
- Behaviour in Crisis Lab, Impact of cumulative stress on the mental health of young people project, Jagiellonian University in Krakow, Krakow, Poland

IPD SHARING:
Plan to Share IPD: Undecided